CLINICAL TRIAL: NCT00823511
Title: The Human Papillomavirus (HPV) Transmission Pilot Study
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-14881; USF IRB 104923
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Human Papillomavirus Infection
Keywords: HPV; Human Papillomavirus Infection; Cervix Uteri; Cancer Control; Risk Assessment, Detection & Intervention; Sexually Transmitted; Neoplasia; Carcinogenesis; Cervix
MeSH Terms: conditions — Papillomavirus Infections; Neoplasms; Carcinogenesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Female Partners: Female partners of HIM Study participants

SUMMARY:
This transmission pilot study is a prospective study to determine feasibility of enrolling female partners into an international transmission study. Companion study to MCC-13930.

DETAILED DESCRIPTION:
We planned to enroll 150 female sexual partners, 75 per year for 2 years, of male study participants in the HPV Infection in Men (HIM) Study. The enrollment period is from June 2006 through May 2008 and participants will be followed through May 2010. At all study visits participants will undergo interviews, a physical exam and laboratory analysis for HPV for a total of 5 clinical visits scheduled every 6 months over 2 years of follow-up. In addition, at each study visit, participants will provide blood for HPV antibody analyses. At enrollment, visit 3 and visit 5 a Pap smear test will be done. At the enrollment visit, study participants will complete a questionnaire designed to assess social and behavioral risk factors for the acquisition of HPV. At each subsequent study visit, participants will be asked to provide updated information to assess changes in risk behaviors such as condom use, relations with new partners, and tobacco use.

ELIGIBILITY:
Inclusion Criteria:

* Female partners of HIM Study participants
* report no abnormal Pap smear during the past 6 months;
* have not had a hysterectomy
* have never been diagnosed with genital warts;
* are not pregnant;
* residents of southern Florida;
* are not and have not been enrolled in an HPV vaccine trial;
* willing to comply with scheduled visits every 6 months for 2 years.

Exclusion Criteria:

* Do not meet the Inclusion Criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female partners of HIM Study participants - Companion study to MCC-13930. Residents of Southern Florida.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2006-10; Primary Completion 2012-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Proportion of men in the HIM study willing to invite their female partner to participate in partner study, proportion of female partners who: a) contact clinic for enrollment in study b) are eligible to participate in the study c) enroll in study. | 2 year accrual period

SECONDARY OUTCOMES:
Proportion of female partners who report being monogamous with the HIM partner, proportion of women that are both HPV sero negative and HPV DNA negative at enrollment, proportion of women who comply with study protocol over 2 years of follow up. | 2 years per participant

CONTACTS AND LOCATIONS:
Overall Officials: Anna Giuliano, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- Moffitt Cancer Center & Research Institute, Tampa, Florida, United States